CLINICAL TRIAL: NCT04287998
Title: Role and Expression of Matrix-remodelling Associated 5 Protein (MXRA5) in Connective Tissue Remodelling of Placenta in Preeclampsia
Brief Title: Role and Expression of MXRA5 in Placental Connective Tissue Remodelling in Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Ahmed Abdelrahman, Principal Investigator, Assiut University
Other Study IDs: MXRA5 in preeclampsia
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Pre-Eclampsia
Keywords: MXRA5; ANXA4; Syndecan1; TIMP1; lead; arsenic
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Placental Tissue samples collection:
  • Placental tissue samples (surgically obtained during the caesarean section from 50 pregnant women) will be selected:
  * 25 PE patients undergoing the caesarean section following confirmation of diagnosis clinically by blood pressure measurement and by urine analysis to detect the proteinuria.
  * 25 control women undergoing the caesarean section. Blood samples. Urinary samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: PE group
- 2: Control group

SUMMARY:
1. To measure the level of expression of MXRA5 and ANXA4 genes in preeclampsia (PE).
2. To detect the effect of heavy metals (lead (Pb) and arsenic (AR)) on these two genes in the pathology of PE.
3. To explore the association of the previous two genes with the heavy metals in link with Phosphoinositide 3-kinases/Protein Kinase B (PI3K/AKT) pathway.
4. To detect Syndecan-1 by immunohistochemical antibodies.
5. To define the role of extracellular matrix remodelling in PE.

DETAILED DESCRIPTION:
* Preeclampsia (PE) is a diverse multisystem syndrome defined as a new onset of hypertension along with evidence of significant multiorgan dysfunction in previously normotensive women 20 weeks of gestation (1)
* The incidence of PE is around 2 - 8 % of pregnancies and it causes about 50,000 deaths worldwide every year (2).
* In Egypt, it complicates 6% - 8% of pregnancies (3).
* Placentation processes include trophoblastic invasion, vascularization of trophoblast to establish and maintain feto-placental vasculature, and subsequent maternal vascular remodeling (4). Extravillous trophoblastic (EVT) cells are crucial for this process (5). If the function of extravillous trophoblast cells is deficient, it can result in PE (6).
* PI3K/AKT pathway plays important roles in placental development and fetal growth (7). PI3K/AKT signaling pathway is important for cell proliferation, migration, invasion and glycolysis/gluconeogenesis (8). AKT can further activate different downstream factors, which plays a predominant role in angiogenesis, vascular permeability and migration (9).
* Matrix metalloproteinase (MMPs) are essential proteases for trophoblast invasion and migration as they promote degrading of the extracellular matrix improving the the cell invasion, while the tissue inhibitors of matrix metalloproteinases (TIMPs) are normal tissue proteins that inhibit the action of MMPs (10).
* Annexin A4 (ANXA4) has been shown to participate in regulation of cellular growth, invasion, and apoptosis. ANXA4 has role in many forms of cancer (11). It was found that ANXA4 expression was downregulated in PE placentas compared with the normal placentas. However, the exact role of ANXA4 in the invasion and survival of trophoblast cells remains less understood.
* ANXA4 binds to the plasma membrane in a Ca2+- dependent manner and regulates its downstream signaling transduction, including phosphoinositide-3-kinase PI3K/AKT signalling (12).
* Matrix-remodelling associated 5 (MXRA5) is a member of the MXRA protein family, participating in cell adhesion and extracellular matrix remodelling (13). This protein is expressed in primates but not in rat or mouse. The function of this protein remains elusive. It resembles the vascular endothelial growth factor (VEGF) receptor and has anti-inflammatory and anti-fibrotic properties (14). Somatic mutations of MXRA5 are found in non-small cell lung cancer and in colorectal cancer (15).
* The expression of MXRA5 was shown to be downregulated in the placentae of PE patients which consequently leads to the inhibition of PI3k/AKT pathway (16).
* As regard that both of ANXA4 and MXRA5 downregulate PI3k/AKT pathway, they are associated to be linked to the pathogenesis of PE.
* Endothelial glycocalyx (EG), the most important protective structure of the endothelium, is an external layer of endothelial cells composed of different proteoglycans (PGs), glycoproteins, glycolipids, and glycosaminoglycans (GAGs). The protective role of EG for endothelium includes for example maintenance of tissue integrity, prevention of leukocytes and platelet adhesion and antithrombotic activity (17). Examples of clinical consequences of EG damage are albuminuria and edema (18).
* Syndecan-1 (SDC-1) is one of the important PGs of EG (19).
* Lead (Pb) is a widespread heavy metal pollutant. Excess Pb in the environment is usually produced via anthropogenic activities, such as mining and untreated sewage irrigation water (20).
* Arsenic (Ar) is a major toxicant in the environment, and a high level of exposure carries an increased risk of cancers and many disorders (21).
* Both of lead and arsenic have been proven to inhibit the PI3K/AKT pathway (22), (23). In this study, lead (Pb) and arsenic (Ar) will be linked to PE through inhibition of PI3K/AKT pathway.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age is >28 weeks.
* Clinically diagnosed PE with blood pressure (≥140/90 mmHg) and proteinuria (≥300mg/dl).
* Healthy pregnant women (age matched control group).

Exclusion Criteria:

* Gestational diabetes.
* Pregestational hypertension (essential hypertension) or proteinuria.
* Systemic illness.
* Vaginal infection.
* Major known fetal or chromosomal anomalies.
* Multiple gestations.
* Intrauterine infections.
* Preterm premature rupture of membranes.
* Sepsis.
* Fever.
* Colitis ulcerosa.
* Crohn's disease.
* Chronic renal disease.
* Rheumatic disease.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: • Placental tissue samples (surgically obtained during the caesarean section from 50 pregnant women) will be selected:
  * 25 PE patients undergoing caesarean section following diagnosis by blood pressure measurement and urine analysis.
  * 25 controls undergoing caesarean section.
  * Placental samples are 4x6 cm in dimension.
  Blood samples:
  Six milliliters of maternal blood was collected in plastic tubes. Urinary samples.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Gene expression level of MXRA5 gene in PE patients and control group | 1 year

SECONDARY OUTCOMES:
Gene expression level of ANXA4 in PE patients and control group. | 1 year
Gene expression level of TIMP1 gene in PE patients and control group. | 1 year
Protein level measurement of phosphorylated AKT(pAKT) in PE patients and control group. | 1 year
Measurement of lead and arsenic level in PE patients and control group. | 1 year